CLINICAL TRIAL: NCT04526210
Title: A Phase 1, Randomized, 2-Period, 2-Sequence, Cross-over Study to Determine the Effect of ALXN1840 on the Metabolism of a CYP2B6 Substrate in Healthy Participants
Brief Title: Study of ALXN1840 on the Metabolism of a CYP2B6 Substrate in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1840-HV-103
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-10

CONDITIONS: Wilson Disease
Keywords: Cytochrome P450; Healthy; ALXN1840
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — tetrathiomolybdate; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will receive bupropion.
  Interventions: Drug: Bupropion Hydrochloride
- Treatment B (Experimental): Participants will receive bupropion with ALXN1840.
  Interventions: Drug: ALXN1840; Drug: Bupropion Hydrochloride

INTERVENTIONS:
Drug: ALXN1840 — ALXN1840 will be administered orally as a single dose as 4 x 15 mg enteric-coated tablets with 240 milliliters of water (fasting), for a total dose of 60 mg.
  Other Names: WTX101; Bis-choline tetrathiomolybdate; Tiomolibdate choline
  Arms: Treatment B
Drug: Bupropion Hydrochloride — Bupropion hydrochloride will be administered orally as a single dose as one 150 milligrams (mg) tablet with 240 milliliters of water (fasting).
  Other Names: Wellbutrin SR 150

SUMMARY:
This is a Phase 1, randomized, 2-period, 2-sequence, cross-over study designed to determine the effect of ALXN1840 on the metabolism of bupropion, a sensitive cytochrome P450 2B6 (CYP2B6) substrate, in healthy male and female participants. The safety and tolerability of ALXN1840 will be determined along with ALXN1840 pharmacokinetics (PK) in plasma as measured via total molybdenum with the coadministration of bupropion.

DETAILED DESCRIPTION:
The study is being conducted as a randomized, 2-period, 2-sequence, cross-over study to determine the effect of a single dose of ALXN1840 (perpetrator) on the single-dose bupropion (victim) kinetics in healthy male and female participants.

The study has a Screening Period (Day -28 to Day -2), two 11-day study periods (Day 1 to Day 11) with a minimum of 14 days between doses of bupropion, and an End of Study Visit (Day 15 ± 2 days) after Period 2 dosing. Participants will report to the clinical research unit on the day prior (Day -1) to both dosing periods. All participants will receive 1 treatment in each study period; treatment order will be defined based on randomization: Treatments A and B.

The time between dosing bupropion alone or in combination with ALXN1840 in each treatment sequence will be a minimum of 14 days.

The PK profile of ALXN1840 and bupropion will be determined by blood sampling following single dose administration.

ELIGIBILITY:
Inclusion Criteria:

* Adequate venous access in the left or right arm to allow the collection of blood samples.
* Body weight ≥ 45 to ≤ 100 kilograms (kg) and body mass index within the range of 18 to < 30 kg/meter squared.
* Willing and able to follow protocol-specified contraception requirements.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of/significant medical history.
* Clinically significant multiple or severe allergies.
* Lymphoma, leukemia, or any malignancy within 5 years.
* Breast cancer within the past 10 years.
* Serum creatinine > upper limit of normal (ULN) of the reference range.
* Alanine aminotransferase, aspartate aminotransferase, or total bilirubin > ULN.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTc > 450 milliseconds (msec) for male participants or > 470 msec for female participants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized to 1 of the two treatment sequences (A-B or B-A) on Day 1 prior to dosing in Period 1. Participants were scheduled to receive a single treatment (A or B) on Day 1 of each treatment period in the crossover design.
Groups:
- Treatment Sequence A-B: Treatment A: Participants received a single oral dose of 1 × 150 milligrams (mg) bupropion hydrochloride (HCl) salt tablet in a fasted state on Day 1 of treatment period 1. Treatment B: Participants received a single oral dose of 1 × 150 mg bupropion HCl salt tablet coadministered with 4 × 15 mg enteric coated (EC) tablets of ALXN1840 in a fasted state on Day 1 of treatment period 2. There was a washout period of 14 days between the 2 treatment periods.
- Treatment Sequence B-A: Treatment B: Participants received a single oral dose of 1 × 150 mg bupropion HCl salt tablet coadministered with 4 × 15 mg EC tablets of ALXN1840 in a fasted state on Day 1 of treatment period 1. Treatment A: Participants received a single oral dose of 1 × 150 mg bupropion HCl salt tablet in a fasted state on Day 1 of treatment period 2. There was a washout period of 14 days between the 2 treatment periods.
Period: Overall Study
Arm/Group | Treatment Sequence A-B | Treatment Sequence B-A
Started | 27 | 27
Received at Least 1 Dose of Stud Drug | 27 (4 participants received Treatment A only.) | 27 (4 participants received Treatment B only.)
Completed | 17 | 20
Not Completed | 10 | 7
Not completed — Sponsor decision | 7 | 5
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least 1 dose of study intervention.
Groups:
- Treatment Sequence A-B: Participants received a single oral dose of 1 × 150 mg bupropion HCl salt tablet in a fasted state on Day 1 of treatment period 1. Treatment B: Participants received a single oral dose of 1 × 150 mg bupropion HCl salt tablet coadministered with 4 × 15 mg EC tablets of ALXN1840 in a fasted state on Day 1 of treatment period 2. There was a washout period of 14 days between the 2 treatment periods.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A-B | Treatment Sequence B-A | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (8.68) | 33.1 (9.22) | 32.3 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 15 | 19 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 4 | 14
  White | 17 | 20 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Bupropion With and Without the Coadministration of ALXN1840
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: Pharmacokinetic (PK) analysis set included all participants who had sufficient plasma samples to have evaluable PK data for bupropion and/or total molybdenum (as a measure of ALXN1840) in plasma. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)/milliliter (mL)
Groups:
- Treatment A: Bupropion HCl: Participants received a single oral dose of 1 × 150 mg bupropion HCl salt tablet in a fasted state on Day 1 of treatment period 1 or 2.
- Treatment B: Bupropion HCl + ALXN1840: Participants received a single oral dose of 1 × 150 mg bupropion HCl salt tablet coadministered with 4 × 15 mg EC tablets of ALXN1840 in a fasted state on Day 1 of treatment period 1 or 2.
Arm/Group | Treatment A: Bupropion HCl | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 37 | 36
nanograms (ng)/milliliter (mL) | 98.64 (31.6) | 98.02 (27.9)
Statistical Analysis 1: Comparison: Treatment A: Bupropion HCl vs Treatment B: Bupropion HCl + ALXN1840; Test type: Other; Geometric least square (LS) mean ratio = 0.980, 90% CI 2-sided [0.9415 to 1.0205]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Last Quantifiable Concentration (AUCt) of Bupropion With and Without the Coadministration of ALXN1840
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: PK analysis set included all participants who had sufficient plasma samples to have evaluable PK data for bupropion and/or total molybdenum (as a measure of ALXN1840) in plasma. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Treatment A: Bupropion HCl | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 37 | 36
hours*ng/mL | 1021 (33.4) | 1010 (31.6)
Statistical Analysis 1: Comparison: Treatment A: Bupropion HCl vs Treatment B: Bupropion HCl + ALXN1840; Test type: Other; Geometric LS mean ratio = 0.978, 90% CI 2-sided [0.9344 to 1.0244]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity (AUCinf) of Bupropion With and Without the Coadministration of ALXN1840
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Treatment A: Bupropion HCl | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 37 | 36
hours*ng/mL | 1049 (32.9) | 1039 (31.3)
Statistical Analysis 1: Comparison: Treatment A: Bupropion HCl vs Treatment B: Bupropion HCl + ALXN1840; Test type: Other; Geometric LS mean ratio = 0.981, 90% CI 2-sided [0.9368 to 1.0269]

4. Secondary Outcome: Cmax of Hydroxybupropion With and Without the Coadministration of ALXN1840
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Bupropion HCl | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 37 | 36
ng/mL | 286.5 (53.8) | 284.3 (53.6)

5. Secondary Outcome: AUCt of Hydroxybupropion With and Without the Coadministration of ALXN1840
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Treatment A: Bupropion HCl | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 37 | 36
hours*ng/mL | 11900 (60.2) | 11560 (55.3)

6. Secondary Outcome: AUCinf of Hydroxybupropion With and Without the Coadministration of ALXN1840
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Treatment A: Bupropion HCl | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 37 | 36
hours*ng/mL | 11960 (59.5) | 11630 (54.8)

7. Secondary Outcome: Cmax of Plasma Total Molybdenum With Coadministration of Bupropion
Description: Plasma total molybdenum was assessed as surrogate measures for ALXN1840 PK following coadministration with bupropion HCl salt tablet (Treatment B) only.
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 46
ng/mL | 325.6 (51.1)

8. Secondary Outcome: AUCt of Plasma Total Molybdenum With Coadministration of Bupropion
Description: as for outcome 7
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 46
hours*ng/mL | 15010 (68.1)

9. Secondary Outcome: AUCinf of Plasma Total Molybdenum With Coadministration of Bupropion
Description: as for outcome 7
Time Frame: Pre-dose (Day 1) up to 336 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 45
hours*ng/mL | 16130 (65.9)

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered with the study drug and which did not necessarily have a causal relationship with the study drug. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A TEAE was defined as any AE that began or worsened on or after the first dose of treatment until the end of study (EOS) or early termination (ET). An AE that occurred during the washout period between drugs was considered treatment emergent to the last drug given. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Day 1 up to Day 15
Population: Safety set included all participants who received at least 1 dose of study intervention.
Measure: Number; unit: participants
Arm/Group | Treatment A: Bupropion HCl | Treatment B: Bupropion HCl + ALXN1840
Number analyzed (Participants) | 50 | 50
participants | 8 | 11

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 15
Description: Safety set included all participants who received at least 1 dose of study intervention.
  All randomized participants except 8 received both assigned doses; 4 participants received only Treatment A and 4 participants received only Treatment B. In total, 50 participants received Treatment A and 50 participants received Treatment B. An AE that occurred during the washout period between drugs was considered treatment emergent to the last drug given.
Arm/Group | Treatment A: Bupropion HCl | Treatment B: Bupropion HCl + ALXN1840
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 8/50 | 11/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Bupropion HCl (N=50) | Treatment B: Bupropion HCl + ALXN1840 (N=50)
Chalazion (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 4
Dizziness (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04526210/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT04526210/SAP_001.pdf